CLINICAL TRIAL: NCT04997239
Title: An Exploratory Clinical Trial to Evaluate the Immunogenicity and Safety of One vs Two Doses of Quadrivalent Influenza Vaccine in Children Aged 3-8 Years Old
Brief Title: A Clinical Trial of Quadrivalent Influenza Vaccine in Children Aged 3-8 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-QINF-4002
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-07

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group ：Vaccine-unprimed subjects with two doses (Experimental): 200 vaccine-unprimed children will receive two doses of quadrivalent influenza vaccine on the immunization schedule of day 0,28.
  Interventions: Biological: Two doses of quadrivalent influenza vaccine
- Experimental Group ：Vaccine-unprimed subjects with one dose (Experimental): 200 vaccine-unprimed children will receive one dose of quadrivalent influenza vaccine.
  Interventions: Biological: One dose of quadrivalent influenza vaccine
- Experimental Group：Vaccine-primed subjects with one dose (Experimental): 200 vaccine-primed children will receive one dose of quadrivalent influenza vaccine.
  Interventions: Biological: One dose of quadrivalent influenza vaccine

INTERVENTIONS:
Biological: Two doses of quadrivalent influenza vaccine — 15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administation is Intramuscular injection into deltoid region.And the immunization schedule is two doses of quadrivalent influenza vaccine on day 0, 28.
  Arms: Experimental Group ：Vaccine-unprimed subjects with two doses
Biological: One dose of quadrivalent influenza vaccine — 15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administation is Intramuscular injection into deltoid region.And the immunization schedule is one dose of quadrivalent influenza vaccine on day 0.
  Arms: Experimental Group ：Vaccine-unprimed subjects with one dose; Experimental Group：Vaccine-primed subjects with one dose

SUMMARY:
This is an open-label, randomized and controlled phase Ⅳ clinical trial of quadrivalent influenza vaccine manufactured by Sinovac Biotech Co. , the purpose of this study is to compare the immunogenicity and safety after 1 dose of quadrivalent influenza vaccine with that of 2 doses in vaccine-unprimed children aged 3-8 years old,to compare the immunogenicity and safety after 1 dose of quadrivalent influenza vaccine in vaccine-unprimed children aged 3-8 years old with that of 1 dose in vaccine-primed children and to compare the immunogenicity and safety after 2 doses of quadrivalent influenza vaccine in vaccine-unprimed children aged 3-8 years old with that of 1 dose in vaccine-primed children.

DETAILED DESCRIPTION:
This study is open-label, randomized and controlled phase Ⅳ clinical trial of quadrivalent influenza vaccine.The purpose of this study is to compare the immunogenicity and safety after 1 dose of quadrivalent influenza vaccine with that of 2 doses in vaccine-unprimed children aged 3-8 years old,to compare the immunogenicity and safety after 1 dose of quadrivalent influenza vaccine in vaccine-unprimed children aged 3-8 years old with that of 1 dose in vaccine-primed children and to compare the immunogenicity and safety after 2 doses of quadrivalent influenza vaccine in vaccine-unprimed children aged 3-8 years old with that of 1 dose in vaccine-primed children.A total of 600 subjects including 400 vaccine-unprimed children and 200 vaccine-primed children will be enrolled,400 vaccine-unprimed children will be randomly divided into two groups in a 1:1 ratio.Subjects in group 1(experimental group 1 ) will receive two doses of quadrivalent influenza vaccine on the immunization schedule of day 0,28 and subjects in group 2 (experimental group 2) will receive one dose of quadrivalent influenza vaccine.200 vaccine-primed children (experimental group 3) will receive one dose of quadrivalent influenza vaccine.

ELIGIBILITY:
vaccine-unprimed children

Inclusion Criteria:

* Healthy children aged 3-8 years;
* The subjects' guardians can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* Received any circulating seasonal influenza vaccine prior to enrollment or had an influenza vaccine schedule during the study;
* Suffering from seasonal influenza in the past 6 moths;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia,functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial. vaccine-primed children

Inclusion Criteria:

* Healthy children aged 3-8 years;
* The subjects' guardians can understand and voluntarily sign the informed consent form;
* Proven legal identity;
* Received at least 1 dose of seasonal influenza vaccine in previous epidemic seasons

Exclusion Criteria:

* Received an seasonal influenza vaccine for the current epidemic season (2020-2021 epidemic season) prior to enrollment, or had an influenza vaccine schedule during the study;
* Suffering from seasonal influenza in the past 6 moths;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index of the seroconversion rate | 28 days after the vaccination of the last dose
  The seroconversion rate of each influenza strain after each dose of quadrivalent influenza vaccine
Immunogenicity index of the seroprotective rate | 28 days after the vaccination of the last dose
  The seroprotective rate of each influenza strain after each dose of quadrivalent influenza vaccine
Immunogenicity index of the GMT | 28 days after the vaccination of the last dose
  The GMT of each influenza strain after each dose of quadrivalent influenza vaccine
Immunogenicity index of the GMI | 28 days after the vaccination of the last dose
  The GMI of each influenza strain after each dose of quadrivalent influenza vaccine
Safety index of the incidence of adverse reactions | From day 0 to day 7 after each dose vaccination
  The incidence of adverse reactions within 0-7 days after each dose
Safety index of the incidence of adverse reactions | From day 0 to day 28 after each dose vaccination
  The incidence of adverse reactions within 0-28 days after each dose
Safety index of the incidence of serious adverse events(SAEs) | From the beginning of the vaccination to 28 days after the whole-schedule vaccination
  The incidence of serious adverse events from the beginning of vaccination to 28 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Huaiyin Center for Disease Control and Prevention, Huai'an, Jiangsu, China